CLINICAL TRIAL: NCT02279238
Title: The Comparison of the 3 Minutes Ramp Walk Test With 6 Minutes Walk Test in Stable Patients After Valve Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PSG Institute of Medical Science and Research (Other)
Collaborators: PSG College of Physiotherapy (Other)
Responsible Party: Principal Investigator, arumugam manivel, Mr. Manivel arumugam, PSG Institute of Medical Science and Research
Other Study IDs: 13/208
Record Dates: First submitted 2014-10-14; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Prosthetic Replacement of Mitral Valve; Abnormality of Aortic Valve
MeSH Terms: interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: cardiac rehabilitation — It is a cross over study in which the participants are assigned for two test simultaneously with washout time of 6 hrs . 5th POD patients are randomly assigned to either 6 minute walk test or 3 minute ramp walk test as first test with 6 hours of rest [Washout time] in between the two test.
  6 MWT : The patient is instructed to walk for a period of 6 minute on a 30 meters Hallway with its extent being demarcated by the placement of 2 cones at the extremes of the Hall.
  3 MRWT : The patient is instructed to walk for a period of 3 minute on a Ramp with an elevation of 30 degree and length of 20 meters with its extent being demarcated by the placement of 2 cones at the extremes of the ramp.
  The data of [HR, SPO2, PSG RPE scale, Distance walked, BP] the participants are collected before, during and after the completion of each lap [according to American Thoracic Society [ATS] protocol].

SUMMARY:
In view of assessing the uphill walking capacity and to provide a functional stress test with better sensitivity the investigators need a short term functional stress test over the gold standard six minute walk test....

To demonstrate the significance of 3 minutes ramp walk test over 6 minutes walk test as a functional stress test.

The investigators hypothesize that the investigators three minutes ramp walk test (3MRWT) will be superior to the existing six minutes level walk test (6MWT) in the measurement of functional capacity of post valve replacement patients.

DETAILED DESCRIPTION:
The patients who have undergone valve replacement surgeries face difficulty in their functional activities especially during climbing stairs, walking uphill.

The six minute level walk test has been a gold standard in the assessment of functional capacity in cardio respiratory conditions like, coronary heart diseases , valvular heart diseases, chronic respiratory illness.

Moreover, six minute walk test has been framed to assess the functional capacity in level walking.so far, no test have been developed to assess the functional capacity of the patients during uphill walking and stair climbing.

Though ramp walking ( uphill walking) can be trained using treadmill, it is not feasible for the indian patients as they are not familiar in the treadmill and their fear may also show variation in the functional assessment.

Hence this study has been proposed..

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* 30 to 65 years
* Patient in step down unit(5th post operative day)
* Aortic and Mitral valve replaced patients

Exclusion Criteria:

* Vitally unstable patients, [pyretic, abnormal BP, SpO₂, X-Ray and pain]
* Any arrthymia
* Orthopaedically disabled patients
* Neurologically impaired patients
* Patients with psychologically impaired

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To find a smallest difference of 70% and a minimal correlation of 40%(r=0.4)between two test , walk distance , vital responses at level of significance of 95% and power of the study 90%, we needed at least 45 patients.to allow for drop outs and missing values,50 patients will be included
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-03 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
The distance walked during the test by the participants | 6 minute level walk & 3 minute Ramp walk
  The variables to be correlated are Distance walked [in meters], heart rate responses, , Saturation Responses

SECONDARY OUTCOMES:
blood pressure before and after test | 6 minute level walk& 3minute Ramp walk
Heart rate before and after test | 6 minute level walk& 3minute Ramp walk
SpO2 % before and after test | 6 minute level walk& 3minute Ramp walk

CONTACTS AND LOCATIONS:
Overall Officials: murugesan PR, MS,Mch,DNB, Study Chair — PSG Institute of Medical Science and Research; manivel arumugam, MPT, Principal Investigator — PSG Institute of Medical Science and Research
Locations (1):
- PSG Hospitals, Coimbatore, Tamil Nadu, India